CLINICAL TRIAL: NCT02338843
Title: A Phase 3, Placebo-Controlled, Randomized, Double-Blind, Multi-Center Study of LJPC-501 in Patients With Catecholamine-Resistant Hypotension (CRH)
Brief Title: A Phase 3 Study of LJPC-501 in Patients With Catecholamine-Resistant Hypotension
Acronym: ATHOS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LJ501-CRH01
Record Dates: First submitted 2015-01-01; First posted 2015-01-14 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-01

CONDITIONS: Catecholamine-resistant Hypotension (CRH); Distributive Shock; High Output Shock; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Angiotensin I; Angiotensin II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LJPC-501 (angiotensin II) (Experimental): Treatment arm
  Interventions: Drug: LJPC-501
- Placebo (0.9% sodium chloride solution) (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LJPC-501 — Treatment arm
  Other Names: angiotensin II
  Arms: LJPC-501 (angiotensin II)
Drug: Placebo — PBO
  Other Names: 0.9% Sodium Chloride Solution USP
  Arms: Placebo (0.9% sodium chloride solution)

SUMMARY:
This is a Phase 3, double-blind, randomized study of LJPC-501 (angiotensin II) in adult patients diagnosed with catecholamine-resistant hypotension (CRH) conducted in multiple centers globally.

DETAILED DESCRIPTION:
Catecholamine-resistant hypotension (CRH) is an often fatal condition resulting from an underlying cause such as septic shock, inflammation due to trauma, or severe drug reactions. When these conditions occur, most patients will respond to either volume expansion or vasopressor treatment. However, some patients will require excessive doses of vasopressors and will be deemed to be resistant.

Angiotensin II is a peptide hormone naturally produced by the body that regulates blood pressure via vasoconstriction and sodium reabsorption. LJPC-501 (angiotensin II) is being developed for the treatment of patients with catecholamine-resistant hypotension (CRH).

This is a multi-site, randomized, double-blind, placebo-controlled study. Adult patients with CRH, who are hospitalized in an ICU setting, may be eligible to participate. Approximately 315 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years of age with CRH, defined as those who require a total sum catecholamine dose of > 0.2 mcg/kg/min for a minimum of 6 hours and a maximum of 48 hours, to maintain a MAP between 55-70 mmHg.
2. Patients are required to have central venous access and an arterial line present, and these are expected to remain present for at least the initial 48 hours of study.
3. Patients are required to have an indwelling urinary catheter present, and it is expected to remain present for at least the initial 48 hours of study.
4. Patients must have received at least 25 mL/kg of crystalloid or colloid equivalent over the previous 24-hour period, and be adequately volume resuscitated in the opinion of the treating investigator.
5. Patients must have clinical features of high-output shock by meeting one of the following criteria.

   1. Central venous oxygen saturation (ScvO2) > 70% (either by oximetry catheter or by central venous blood gas) and central venous pressure (CVP) > 8 mmHg.

      OR
   2. Cardiac Index (CI) > 2.3 L/min/1.73 m2. Patient must meet 5a or 5b to be eligible.
6. Patient or legal surrogate is willing and able to provide written informed consent and comply with all protocol requirements.

Exclusion Criteria:

1. Patients who are < 18 years of age.
2. Any patient with burns covering > 20% of total body surface area (TBSA).
3. Patients with a Cardiovascular (CV) SOFA score ≤ 3.
4. Patients diagnosed with acute occlusive coronary syndrome requiring intervention.
5. Patients on veno-arterial (VA) ECMO.
6. Patients who have been on ECMO for less than 12 hours.
7. Patients in liver failure with a Model for End-Stage Liver Disease (MELD) score of ≥ 30.
8. Patients with a history of asthma or who are currently experiencing bronchospasm requiring the use of inhaled bronchodilators, if not mechanically ventilated.
9. Patients with acute mesenteric ischemia or a history of mesenteric ischemic.
10. Patients with a history of, presence of, or highly-suspected of having an aortic dissection or abdominal aortic aneurysm.
11. Patients requiring more than 500 mg daily of hydrocortisone or equivalent glucocorticoid medication as a standing dose.
12. Patients with Raynaud's phenomenon, systemic sclerosis or vasospastic disease.
13. Patients with an expected lifespan of < 12 hours.
14. Patients with active bleeding AND an anticipated need (within 48 hours of initiation of the study) for transfusion of > 4 units of packed red blood cells.
15. Patients with active bleeding AND hemoglobin < 7g/dL or any other condition that would contraindicate serial blood sampling.
16. Patients with an absolute neutrophil count (ANC) of < 1000 cells/mm3.
17. Patients with a known allergy to mannitol.
18. Patients who are current participating in another interventional clinical trial.
19. Patients who are known to be pregnant at the time of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12-01 (Actual); Study Completion 2017-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George F Tidmarsh, MD, PhD, Study Director — La Jolla Pharmaceutical Company
Locations (115):
- United States (52):
  - Pulmonary Associates of Mobile, PC, Mobile, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles County + University of Southern California Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - University of California, Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Joseph M. Still Research Foundation, Inc., Augusta, Georgia
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Methodist Hospital, Indiana University Health Physicians, Indianapolis, Indiana
  - Kentucky Lung Clinic, Hazard, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Paul Regions Hospital, Saint Paul, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Sunrise Hospital/eStudySite, Las Vegas, Nevada
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Rutgers Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Montefiore Medical Center, Weiler Division, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses Cone Health, Greensboro, North Carolina
  - Wesley Long Hospital, Greensboro, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic - Fairview Hospital, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Erlanger Hospital, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Baylor University, Dallas, Texas
  - John Peter Smith Hospital - JPS Health Network, Fort Worth, Texas
  - U.S. Army Military Medical Center, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Australia (18):
  - Canberra Hospital, Garran, Australian Capital Territory
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - St. Vincent's Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
- Belgium (5):
  - UZ Antwerpen, Antwerp
  - Brugmann University Hospital, Brussels
  - Erasme University Hospital, Brussels
  - UZ Brussel, Brussels
  - UZ Gent, Ghent
- Canada (10):
  - South Health Campus & Rockyview General Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (4):
  - Jean Minjoz Hospital, Besançon
  - Hospital Roger Salengro, CHRU de Lille, Lille
  - CHU Nice, Nice
  - Bordeaux Hospital University Center, Pessac
- Germany (2):
  - University Medical Center, Berlin, Berlin
  - University Hospital Münster, Münster
- New Zealand (3):
  - Auckland City Hospital, Grafton, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - Wellington Hospital, Newtown, Wellington Region
- Bern University Hospital, Bern, Switzerland
- United Kingdom (16):
  - Southampton General Hospital, Southampton, Hampshire
  - Norfolk and Norwich University Hospitals, Norwich, Norfolk
  - Sunderland Royal Hospital, Sunderland, Tyne and Wear
  - Birmingham Heartlands Hospital, Birmingham, West Midlands
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Hull Royal Infirmary, Hull
  - Royal London Hospital, London
  - St. Thomas Hospital, London
  - St. George's University Hospital, London
  - Charing Cross Hospital, London
  - Hammersmith Hospital, London
  - Royal Liverpool Hospital, Merseyside
  - Northampton General Hospital, Northampton
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Leisman DE, Wieruszewski PM, Busse LW, Chawla LS, Hibbert KA, Handisides DR, Khanna AK, Ostermann M, McCurdy MT, Adams CD, Hodges TN, Bellomo R; ATHOS-3 Investigators. An index of the initial blood pressure response to angiotensin II treatment and its association with clinical outcomes in vasodilatory shock. Crit Care. 2025 Feb 19;29(1):81. doi: 10.1186/s13054-025-05311-z. PMID 39972379
- [Derived] Leisman DE, Handisides DR, Busse LW, Chappell MC, Chawla LS, Filbin MR, Goldberg MB, Ham KR, Khanna AK, Ostermann M, McCurdy MT, Adams CD, Hodges TN, Bellomo R; ATHOS-3 Investigators. ACE inhibitors and angiotensin receptor blockers differentially alter the response to angiotensin II treatment in vasodilatory shock. Crit Care. 2024 Apr 18;28(1):130. doi: 10.1186/s13054-024-04910-6. PMID 38637829
- [Derived] Leisman DE, Handisides DR, Chawla LS, Albertson TE, Busse LW, Boldt DW, Deane AM, Gong MN, Ham KR, Khanna AK, Ostermann M, McCurdy MT, Thompson BT, Tumlin JS, Adams CD, Hodges TN, Bellomo R. Angiotensin II treatment is associated with improved oxygenation in ARDS patients with refractory vasodilatory shock. Ann Intensive Care. 2023 Dec 16;13(1):128. doi: 10.1186/s13613-023-01227-5. PMID 38103056
- [Derived] Wieruszewski PM, Bellomo R, Busse LW, Ham KR, Zarbock A, Khanna AK, Deane AM, Ostermann M, Wunderink RG, Boldt DW, Kroll S, Greenfeld CR, Hodges T, Chow JH; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Initiating angiotensin II at lower vasopressor doses in vasodilatory shock: an exploratory post-hoc analysis of the ATHOS-3 clinical trial. Crit Care. 2023 May 5;27(1):175. doi: 10.1186/s13054-023-04446-1. PMID 37147690
- [Derived] Bellomo R, Forni LG, Busse LW, McCurdy MT, Ham KR, Boldt DW, Hastbacka J, Khanna AK, Albertson TE, Tumlin J, Storey K, Handisides D, Tidmarsh GF, Chawla LS, Ostermann M. Renin and Survival in Patients Given Angiotensin II for Catecholamine-Resistant Vasodilatory Shock. A Clinical Trial. Am J Respir Crit Care Med. 2020 Nov 1;202(9):1253-1261. doi: 10.1164/rccm.201911-2172OC. PMID 32609011
- [Derived] Bellomo R, Wunderink RG, Szerlip H, English SW, Busse LW, Deane AM, Khanna AK, McCurdy MT, Ostermann M, Young PJ, Handisides DR, Chawla LS, Tidmarsh GF, Albertson TE. Angiotensin I and angiotensin II concentrations and their ratio in catecholamine-resistant vasodilatory shock. Crit Care. 2020 Feb 6;24(1):43. doi: 10.1186/s13054-020-2733-x. PMID 32028998
- [Derived] Senatore F, Jagadeesh G, Rose M, Pillai VC, Hariharan S, Liu Q, McDowell TY, Sapru MK, Southworth MR, Stockbridge N. FDA Approval of Angiotensin II for the Treatment of Hypotension in Adults with Distributive Shock. Am J Cardiovasc Drugs. 2019 Feb;19(1):11-20. doi: 10.1007/s40256-018-0297-9. PMID 30144016
- [Derived] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Derived] Schmull S, Wang Z, Gao L, Lv J, Li J, Xue S. Angiotensins and Their Receptors in Cardiac and Vascular Injury. Curr Hypertens Rev. 2016;12(3):170-180. doi: 10.2174/1573402112666160302101545. PMID 26931475

RESULTS

PARTICIPANT FLOW:
Groups:
- LJPC-501 (Angiotensin II): Treatment arm Injection for Intravenous Infusion
- Placebo (0.9% Sodium Chloride Solution): Placebo arm Volume matched saline administered via intravenous infusion
Period: Overall Study
Arm/Group | LJPC-501 (Angiotensin II) | Placebo (0.9% Sodium Chloride Solution)
Started (Discrepancy between enrollment and started numbers due to 23 pts who enrolled but were not treated.) | 163 | 158
Completed | 119 | 100
Not Completed | 44 | 58
Not completed — Adverse Event | 2 | 1
Not completed — Death | 40 | 53
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Subject Recovered | 0 | 2
Not completed — Discontinued prior to randomizat | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LJPC-501 (Angiotensin II) | Placebo (0.9% Sodium Chloride Solution) | Total
Number analyzed (Participants) | 163 | 158 | 321
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [52 to 75] | 65 [53 to 75] | 64 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 55 | 126
  Male | 92 | 103 | 195
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 4 | 5 | 9
  Canada | 26 | 10 | 36
  Belgium | 0 | 1 | 1
  United States | 90 | 110 | 200
  Finland | 5 | 2 | 7
  United Kingdom | 9 | 9 | 18
  Australia | 24 | 19 | 43
  France | 5 | 1 | 6
  Germany | 0 | 1 | 1
Body Mass Index (BMI) [Count of Participants; unit: Participants] — Population: BMI could not be calculated for two patients in the treatment group and three patients in the placebo group.
  Participants
    BMI ≥ 30: number analyzed (Participants) | 161 | 155 | 316
    BMI ≥ 30 | 69 | 71 | 140
    BMI < 30: number analyzed (Participants) | 161 | 155 | 316
    BMI < 30 | 92 | 84 | 176
Mean Arterial Pressure (MAP) [Median (Inter-Quartile Range); unit: mmHg] | 66.3 [63.7 to 69.0] | 66.3 [63.0 to 68.3] | 66.3 [63.7 to 68.7]
APACHE II Score [Median (Inter-Quartile Range); unit: points] — The Acute Physiology and Chronic Health Evaluation (APACHE II) is a severity score and mortality estimation tool developed from a large sample of ICU patients in the United States. The APACHE II score is made of 12 physiological variables and 2 disease-related variables. The APACHE II score ranges from 0 to 71 points, with higher scores correlating to worse outcomes.
  points | 27 [22 to 33] | 29 [22 to 34] | 28 [22 to 33]
Vasopressor Dose [Median (Inter-Quartile Range); unit: mcg/kg/min] | 0.33 [0.23 to 0.56] | 0.34 [0.23 to 0.56] | 0.34 [0.23 to 0.56]
Cause of Shock [Count of Participants; unit: Participants]
  Sepsis | 127 | 132 | 259
  Other, potentially sepsis | 20 | 11 | 31
  Pancreatitis | 0 | 2 | 2
  Vasoplegia | 10 | 9 | 19
  Other | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: An Increased MAP, Defined as Achievement of a Day 1 MAP at 3 Hours Following the Initiation of Study Drug, of ≥ 75 mmHg OR a 10 mmHg Increase in Baseline MAP
Description: Response with respect to mean arterial pressure (MAP) at hour 3 after the start of infusion was defined as an increase from baseline of at least 10 mm Hg or an increase to at least 75 mm Hg, without an increase in the dose of background vasopressors.
Time Frame: Hour 3
Measure: Count of Participants; unit: Participants
Arm/Group | LJPC-501 (Angiotensin II) | Placebo (0.9% Sodium Chloride Solution)
Number analyzed (Participants) | 163 | 158
Participants | 114 | 37
Statistical Analysis 1: Comparison: LJPC-501 (Angiotensin II) vs Placebo (0.9% Sodium Chloride Solution); Test type: Superiority; p < 0.001, Regression, Logistic; Stratified logistic regression model. Adjusted by baseline MAP and APACHE II, vasopressin use and average NED 6 hours prior to randomization; Odds Ratio (OR) = 7.95, 95% CI 2-sided [4.76 to 13.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study drug initiation through Day 28.
Arm/Group | LJPC-501 (Angiotensin II) | Placebo (0.9% Sodium Chloride Solution)
All-Cause Mortality (participants affected / at risk) | 75/163 | 85/158
Serious Adverse Events (participants affected / at risk) | 99/163 | 106/158
Other Adverse Events (participants affected / at risk) | 110/163 | 108/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LJPC-501 (Angiotensin II) (N=163) | Placebo (0.9% Sodium Chloride Solution) (N=158)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cardiac valve vegetation (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 18 (18) | 10 (10)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mental status change (Psychiatric disorders) | 1 (1) | 0 (0)
Brain hypoxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of conciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Toxic leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 5 (5)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 7 (10) | 9 (10)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 4 (4)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 5 (5) | 3 (3)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0)
Distributive shock (Vascular disorders) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 5 (5) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 5 (5) | 3 (3)
Shock (Vascular disorders) | 3 (3) | 3 (3)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (11)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal mucosal exfoliation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic vascular thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 25 (25) | 23 (23)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (2) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LJPC-501 (Angiotensin II) (N=163) | Placebo (0.9% Sodium Chloride Solution) (N=158)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15) | 10 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (14) | 10 (10)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 11 (11)
Agitation (Psychiatric disorders) | 6 (6) | 8 (8)
Delirium (Psychiatric disorders) | 9 (9) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 17 (18) | 16 (18)
Bradycardia (Cardiac disorders) | 6 (6) | 9 (9)
Hypertension (Vascular disorders) | 9 (11) | 9 (9)
Hypotension (Vascular disorders) | 13 (16) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All investigators were restricted from publishing individual papers until the study-wide publication was published. After this time, investigator restrictions varied by institution.